CLINICAL TRIAL: NCT00739921
Title: PCR Analysis of Nasal Polyps for Fungal DNA
Brief Title: The Polymerase Chain Reaction (PCR) Analysis of Nasal Polyps for Fungal DNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H9272-26987-05
Record Dates: First submitted 2008-08-19; First posted 2008-08-22 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Sinusitis; Nasal Polyps
Keywords: PCR Analysis; Allergic fungal sinusitis; Chronic rhinosinusitis; Nasal Polyps
MeSH Terms: conditions — Sinusitis; Nasal Polyps; Allergic Fungal Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients with sinusitis compared to patients without.
  To find out if any specific type of fungus or mold is correlated with chronic sinus disease. The study will add new information about the different types of fungus and mold found in the human nose.
  Interventions: Procedure: Nasal swab under endoscopic guidance

INTERVENTIONS:
Procedure: Nasal swab under endoscopic guidance — After the application of pontocaine and neosynephrine spray, the following will be done:
  * A small sponge applicator will be used to swab the inside of your mouth for saliva collection
  * A blood sample (6cc - one tube) will be collected
  * A small brush applicator called a cytology brush and an instrument called an endoscope will be used to swab the inside of your nose (middle meatus)
  * Subjects will be asked to complete 2 standard quality of life questionnaires regarding how much your symptoms bother you
  * You will be asked to bring in a vacuum cleaner bag from home at a follow-up appointment which will be swabbed as well
  The samples will be refrigerated and analyzed using PCR to detect and speciate fungus.

SUMMARY:
The objective of this study is to determine whether the amount or type of fungal DNA present in the nose and home environment can be correlated with the outcomes of the following quality of life (QOL) instruments: Medical Outcomes Study 36-item Short Form (SF-36) and the Sino-Nasal Outcomes Study - 20 Questions (SNOT-20).

DETAILED DESCRIPTION:
The objective of this study is to determine whether the amount or type of fungal DNA present in the nose and home environment can be correlated with the outcomes of the following quality of life (QOL) instruments: Medical Outcomes Study 36-item Short Form (SF-36) and the Sino-Nasal Outcomes Study - 20 Questions (SNOT-20).

The study design involves case control Polymerase Chain reaction (PCR) analysis of nasal mucosal swabs, saliva swabs, blood serum, and home vacuum cleaner bags in patients with sinusitis and normal controls.

The hypothesis is that the quantity and type of fungal DNA present in the nose and home environment are directly correlated with quality of life. Our research aims to both quantify the amount of fungi present in the nasal mucosa as well as to measure the severity of the patient's chronic rhinosinusitis (CRS) as a function of SNOT-20 and SF-36 outcomes questionnaires. We hypothesize that the amount and type of fungi present in the nose and home environment will correlate with the severity of the patients' symptoms of CRS.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with no sinus disease and subjects with chronic rhinosinusitis.

Exclusion Criteria:

* Immunocompromise
* Pregnancy
* Minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2006-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Quality of life (QOL) instruments: Medical Outcomes Study 36-Item Short Form (SF-36) and the Sino-Nasal Outcomes Study- 20 questions (SNOT-20). | During the course of outpatient visit

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Murr, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, Dept of Otolaryngology-HNS, San Francisco, California, United States

REFERENCES:
- [Background] Catten MD, Murr AH, Goldstein JA, Mhatre AN, Lalwani AK. Detection of fungi in the nasal mucosa using polymerase chain reaction. Laryngoscope. 2001 Mar;111(3):399-403. doi: 10.1097/00005537-200103000-00006. PMID 11224767
- [Background] Scheuller MC, Murr AH, Goldberg AN, Mhatre AN, Lalwani AK. Quantitative analysis of fungal DNA in chronic rhinosinusitis. Laryngoscope. 2004 Mar;114(3):467-71. doi: 10.1097/00005537-200403000-00015. PMID 15091220
- [Background] Vesper SJ, Varma M, Wymer LJ, Dearborn DG, Sobolewski J, Haugland RA. Quantitative polymerase chain reaction analysis of fungi in dust from homes of infants who developed idiopathic pulmonary hemorrhaging. J Occup Environ Med. 2004 Jun;46(6):596-601. doi: 10.1097/01.jom.0000128160.17144.6e. PMID 15213523